CLINICAL TRIAL: NCT02220686
Title: Vascular Physician Offer and Report (VAPOR) Trial
Acronym: VAPOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Society for Vascular Surgery (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D14197
Record Dates: First submitted 2014-08-14; First posted 2014-08-20 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Peripheral Artery Disease (PAD)
Keywords: VAPOR; smoking cessation; PAD
MeSH Terms: conditions — Peripheral Arterial Disease; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Offer and Report Protocol (Experimental): Physician advice to stop smoking, referral to state Quitline, and physician considers prescribing nicotine replacement therapy.
  Interventions: Behavioral: Offer and Report Protocol
- Usual Care (No Intervention): Physician will follow their institution's standard of care for smoking cessation.

INTERVENTIONS:
Behavioral: Offer and Report Protocol — Physician advice to stop smoking, referral to state Quitline, and physician considers prescribing nicotine replacement therapy.
  Arms: Offer and Report Protocol

SUMMARY:
The purpose of the study is to see if vascular physicians (your provider) using a combination of proven smoking cessation tools in an organized way can help vascular patients quit smoking better than usual.

The doctors where you are being treated have been chosen to either provide:

the combination therapy of giving you advice, considering prescribing medications to help you quit smoking, and referring you to a phone quitline, or to continue their usual smoking cessation practices (which may include all, some, or none of the treatments above).

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Current smoker
* Plan to have a Vascular Quality Initiative (VQI) procedure in > 7 days

Exclusion Criteria:

* Pregnant Women, Fetuses and Neonates
* Children
* People with impaired decision-making capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of the "Offer and Report" protocol for change in smoking status from Baseline Visit to 3 Month Visit | Change in smoking status from Baseline Visit to 3 Month Visit
  To assess the efficacy of the "Offer and Report" protocol (standardized (1) "very brief advice," (2) referral to telephone-based smoking cessation counseling, and (3) consideration of prescribing nicotine replacement therapy (NRT)) as compared to usual smoking cessation care by vascular physicians in biochemically-validated 3 month smoking cessation rates. A questionnaire will be completed by the patient at the Baseline visit and another questionnaire will be completed at the 3 month visit to assess the change in smoking status.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Goodney, MD, MS, Principal Investigator — Dartmouth-Hitchcock Medical Center; Alik Farber, MD, Principal Investigator — Boston Medical Center
Locations (8):
- United States (8):
  - UF Health, Gainesville, Florida
  - Northwestern Memorial, Chicago, Illinois
  - University Health, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - UMASS Memorial Medical Center, Worcester, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Roper Hospital, Charleston, South Carolina
  - University of Utah Hospital, Salt Lake City, Utah

REFERENCES:
- [Derived] Spangler EL, Brooke BS, Beck AW, Hoel A, Farber A, Goodney PP; VAPOR Trial Investigators. Design and initial enrollment in the Vascular Physicians Offer and Report (VAPOR) trial. J Vasc Surg. 2016 Apr;63(4):1121-5.e2. doi: 10.1016/j.jvs.2015.12.026. PMID 27016862